CLINICAL TRIAL: NCT05784753
Title: HEART (Heart Failure Exercise and Resistance Training) Camp Connect: Promoting Adherence to Exercise in Adults With Heart Failure With Preserved Ejection Fraction
Brief Title: HEART Camp Connect -Promoting Exercise in Adults With Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0040-23-FB
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: exercise training; patient adherence; coaching
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Participants will be randomized following a 2-2-1 (HEART Camp Connect - HEART Camp - Enhanced Usual Care) scheme to fully examine comparative effects between virtual and in-person treatment groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded study personnel will participate in all data collection time points, meeting with participants at four time points during the study and confirming completeness of questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HEART Camp (Experimental): Participants in the HEART Camp group will be provided paid, in-person access to the medical fitness center and in-person coaching by a trained coach.
  Interventions: Behavioral: HEART Camp
- HEART Camp Connect (Experimental): Participants in the HEART Camp Connect group will be provided paid, virtual access to the medical fitness center and virtual coaching by a trained coach via videoconference. Participants will also receive automated, asynchronous motivational electronic messaging if they are below the weekly adherence threshold.
  Interventions: Behavioral: HEART Camp Connect
- Enhanced Usual Care (No Intervention): Participants in the Enhanced Usual Care group will be provided paid virtual access to the medical fitness center and virtual availability of the medical fitness center staff and study personnel for participant-initiated questions.

INTERVENTIONS:
Behavioral: HEART Camp — Participants will meet with an in-person coach at the medical fitness center: Months 1-3 weekly for 30 minutes; Months 4-12 every other week for 15 minutes (on alternate weeks, participants will attend a 1-hour group-based exercise training and coaching).
  Arms: HEART Camp
Behavioral: HEART Camp Connect — Participants will meet with a virtual coach from the medical fitness center via videoconferencing: Months 1-3 weekly for 30 minutes; Months 4-12 every other week for 15 minutes (on alternate weeks, participants will attend a virtual 1-hour group-based exercise training and coaching session via videoconferencing).
  Arms: HEART Camp Connect

SUMMARY:
The goal of this study is to learn more about patients with heart failure with preserved ejection fraction (HFpEF) and exercise. Investigators want to see if meeting with a coach in person or by video conference will help these patients exercise, feel better, and change markers in their blood. Participants will be randomly placed in one of three groups for 18 months. All groups will have access to a fitness center and be given a watch and heart rate monitor to wear during exercise. The usual care group (control group) will have access to exercise videos via the medical fitness center and will not meet with a coach. The HEART Camp group will exercise and meet with their coach in-person at the medical fitness center. The HEART Camp Connect group will have access to exercise videos via the medical fitness center and will meet with their coach via videoconferencing. All participants will take part in an exercise test and study training prior to being randomized. At four data collection time points, participants will wear an activity monitor for 7 days each, have their blood drawn, and answer questions related to heart failure and exercise. Participants will also wear a heart rate monitor when they exercise and fill out a daily exercise diary.

DETAILED DESCRIPTION:
The overall objectives for this study are to: (a) test the efficacy of virtual and in-person exercise interventions to promote long-term adherence to exercise; (b) determine a benchmark of exercise minutes that reaches a minimal clinically important difference in heart failure related health status and drives improvements in physical function, inflammatory markers, and patient-reported outcomes; (c) identify interventional mechanisms, interim clinical events and prognostic indicators of heart failure with preserved ejection fraction (HFpEF) that mediate adherence; (d) assess delivery method and related cost of the intervention to support translation and scalability. To meet these objectives, investigators propose a three-group, 2-2-1 randomized repeated measures experimental design with 4 data collection points [baseline, 6, 12, and 18 months to compare HEART Camp, HEART Camp Connect, and virtual enhanced usual care (EUC).

This study begins with the cardiopulmonary exercise testing (CPET) . The CPET is used to develop an exercise prescription and ensure participant safety and readiness for exercise. Participants who have completed a CPET within 6 months of enrollment with no changes in medications will not repeat the test. Any participants who exhibit potential safety concerns during CPET (e.g. cardiac arrhythmias, balance instability) will be evaluated by a trained providers, prior to continuing in the study. Those deemed unsafe to exercise will be withdrawn. After the CPET, participants will take part in the run-in period with 3 monitored sessions in cardiac rehabilitation and study orientation. All participants will be oriented during a one-time in-person training to familiarize them with the 1) Either in-person Engage center or Engage virtual platform via the HEART Camp You Tube channel; 2) All monitoring devices (Polar watch and Polar heart rate monitor, Actigraph, rating of perceived exertion scale, and exercise diary); and 3) Private HEART Camp You Tube channel where they can view investigator-developed educational videos specific to HFpEF and virtual exercise content. Participants who do not have a smart device with internet capability or have an insufficient data plan will be given a tablet with a wireless data plan for study use.

After randomization, participants in the intervention groups (HEART Camp Connect and HEART Camp) meet with a coach for the first 12 months of the study. The HEART Camp group will meet in-person at the medical fitness center with their coach. The HEART Camp Connect group will meet virtually, over videoconference. To improve the scalability of this intervention, investigators will taper coaching sessions according to the following schedule: Months 1-3 weekly, 1-on-1 coaching for 30 minutes; Months 4-12 1-on-1 coaching is reduced to 15 minute sessions every other week. On alternate weeks, participants will attend a 1-hour group-based exercise training and coaching. During these sessions, the coach will meet with 4-6 participants at once. One half of the class will be an exercise training session and the other half will be a question/answer session for participants to talk to the coach and each other about strategies for exercise. After 12 months, coaching (both intervention groups) and motivational messages (HEART Camp Connect only) will stop and participants will be expected to self-regulate exercise in months 13-18.

Participants will be asked to build up to 150 minutes of moderate-intensity exercise weekly. During exercise sessions, participants will be asked to wear their study-provided watch and heart rate monitor and keep a daily exercise diary.

Participants will meet with research personnel at 4 times during the study for data collection including where they will have their blood drawn and complete a 6 minute walk test. At these data collection time points, participants will also wear an activity monitor for 7 days/nights and complete surveys related to their heart failure and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with an ejection fraction greater than or equal to 50
* Echocardiogram in prior 24 months
* Stable pharmacologic therapy in the past 30 days
* Any of the following evidence to confirm HFpEF - Score< 6 on Heavy Hypertensive Atrial Fibrillation, Pulmonary Hypertension, Elder, Filling Pressure algorithm, invasive hemodynamic evidence of HFpEF(i.e., elevated pulmonary wedge pressure), or a confirmed clinical diagnosis of HFpEF

Exclusion Criteria:

* Life-limiting illness precluding study completion
* Clinical evidence of decompensated heart failure
* Unstable angina or marked shortness of breath on exertion at less than 2 metabolic equivalents
* Myocardial infarction, coronary artery bypass graft, or biventricular pacemaker in prior 6 weeks
* Orthopedic or neuromuscular disorders preventing aerobic exercise
* Cardiopulmonary exercise test results that preclude safe exercise
* Unwilling/unable to complete pre-randomization procedures
* Pregnancy
* Implantable cardioverter defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Exercise Adherence | 6 months
  Adherence is measured as weekly minutes of moderate intensity exercise as measured by a watch and heart rate sensor.
Exercise Adherence | 12 months
  Adherence is measured as weekly minutes of moderate intensity exercise as measured by a watch and heart rate sensor.
Exercise Adherence | 18 months
  Adherence is measured as weekly minutes of moderate intensity exercise as measured by a watch and heart rate sensor.

SECONDARY OUTCOMES:
HF-related Health Status | Baseline
  Scores on the Kansas City Cardiomyopathy Questionnaire, assessing the domains of physical limitations, HF symptoms, quality of life, social impact of HF, and self efficacy. A 23-item questionnaire where scores are generated for each domain and scaled from 0-100, with 0 denoting the worst and 100 the best possible status.
HF-related Health Status | 6 months
  Scores on the Kansas City Cardiomyopathy Questionnaire, assessing the domains of physical limitations, HF symptoms, quality of life, social impact of HF, and self efficacy. A 23-item questionnaire where scores are generated for each domain and scaled from 0-100, with 0 denoting the worst and 100 the best possible status.
HF-related Health Status | 12 months
  Scores on the Kansas City Cardiomyopathy Questionnaire, assessing the domains of physical limitations, HF symptoms, quality of life, social impact of HF, and self efficacy. A 23-item questionnaire where scores are generated for each domain and scaled from 0-100, with 0 denoting the worst and 100 the best possible status.
HF-related Health Status | 18 months
  Scores on the Kansas City Cardiomyopathy Questionnaire, assessing the domains of physical limitations, HF symptoms, quality of life, social impact of HF, and self efficacy. A 23-item questionnaire where scores are generated for each domain and scaled from 0-100, with 0 denoting the worst and 100 the best possible status.
Physical Function | Baseline
  Physical function will be measured by distance in meters completed on the 6 minute walk test.
Physical Function | 6 months
  Physical function will be measured by distance in meters completed on the 6 minute walk test.
Physical Function | 12 months
  Physical function will be measured by distance in meters completed on the 6 minute walk test.
Physical Function | 18 months
  Physical function will be measured by distance in meters completed on the 6 minute walk test.
Physical Activity | Baseline
  Physical activity will be assessed based on data gathered from participants wearing an accelerometer for 7 days/nights.
Physical Activity | 6 months
  Physical activity will be assessed based on data gathered from participants wearing an accelerometer for 7 days/nights.
Physical Activity | 12 months
  Physical activity will be assessed based on data gathered from participants wearing an accelerometer for 7 days/nights.
Physical Activity | 18 months
  Physical activity will be assessed based on data gathered from participants wearing an accelerometer for 7 days/nights.
Dyspnea Severity | Baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS)-Dyspnea Severity 10a, assessing severity of shortness of breath in response to different activities over the prior 7-day period. 10 items are assessed on a 4-point Likert scale with raw scores ranging from 0-30. Higher scores indicate greater perceived dyspnea.
Dyspnea Severity | 6 months
  Patient-Reported Outcomes Measurement Information System (PROMIS)-Dyspnea Severity 10a, assessing severity of shortness of breath in response to different activities over the prior 7-day period. 10 items are assessed on a 4-point Likert scale with raw scores ranging from 0-30. Higher scores indicate greater perceived dyspnea.
Dyspnea Severity | 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS)-Dyspnea Severity 10a, assessing severity of shortness of breath in response to different activities over the prior 7-day period. 10 items are assessed on a 4-point Likert scale with raw scores ranging from 0-30. Higher scores indicate greater perceived dyspnea.
Dyspnea Severity | 18 months
  Patient-Reported Outcomes Measurement Information System (PROMIS)-Dyspnea Severity 10a, assessing severity of shortness of breath in response to different activities over the prior 7-day period. 10 items are assessed on a 4-point Likert scale with raw scores ranging from 0-30. Higher scores indicate greater perceived dyspnea.
Global Symptoms | Baseline
  PROMIS-29 Profile v2.1 assessing physical function, anxiety, depression, fatigue, sleep disturbances, satisfaction with social role, pain impact, and pain intensity. Pain intensity is assessed using a single 0-10 numeric rating, The 7 health domains are measured using 4 items per domain that are assessed on a 5-point Likert scale. Each domain is scored separately with raw scores ranging from 4-20, higher scores indicate worse symptomatology.
Global Symptoms | 6 months
  PROMIS-29 Profile v2.1 assessing physical function, anxiety, depression, fatigue, sleep disturbances, satisfaction with social role, pain impact, and pain intensity. Pain intensity is assessed using a single 0-10 numeric rating, The 7 health domains are measured using 4 items per domain that are assessed on a 5-point Likert scale. Each domain is scored separately with raw scores ranging from 4-20, higher scores indicate worse symptomatology.
Global Symptoms | 12 months
  PROMIS-29 Profile v2.1 assessing physical function, anxiety, depression, fatigue, sleep disturbances, satisfaction with social role, pain impact, and pain intensity. Pain intensity is assessed using a single 0-10 numeric rating, The 7 health domains are measured using 4 items per domain that are assessed on a 5-point Likert scale. Each domain is scored separately with raw scores ranging from 4-20, higher scores indicate worse symptomatology.
Global Symptoms | 18 months
  PROMIS-29 Profile v2.1 assessing physical function, anxiety, depression, fatigue, sleep disturbances, satisfaction with social role, pain impact, and pain intensity. Pain intensity is assessed using a single 0-10 numeric rating, The 7 health domains are measured using 4 items per domain that are assessed on a 5-point Likert scale. Each domain is scored separately with raw scores ranging from 4-20, higher scores indicate worse symptomatology.
Health-related Quality of Life | Baseline
  Euro Qual (EQ)-5 Dimension, assessing the five dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 5 items are assessed on a 5-point Likert scale and a summary index with a maximum score of 1 is derived from the 5 dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state.
Health-related Quality of Life | 6 months
  Euro Qual (EQ)-5 Dimension, assessing the five dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 5 items are assessed on a 5-point Likert scale and a summary index with a maximum score of 1 is derived from the 5 dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state.
Health-related Quality of Life | 12 months
  Euro Qual (EQ)-5 Dimension, assessing the five dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 5 items are assessed on a 5-point Likert scale and a summary index with a maximum score of 1 is derived from the 5 dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state.
Health-related Quality of Life | 18 months
  Euro Qual (EQ)-5 Dimension, assessing the five dimensions of mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 5 items are assessed on a 5-point Likert scale and a summary index with a maximum score of 1 is derived from the 5 dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state.
Health Status | Baseline
  Euro Qual (EQ)-Visual Analog Scale, Participants rate their perceived health status on a scale of 0-100 with 0 indicating the worst imaginable health state and 100 indicating the best imaginable health state
Health Status | 6 months
  Euro Qual (EQ)-Visual Analog Scale, Participants rate their perceived health status on a scale of 0-100 with 0 indicating the worst imaginable health state and 100 indicating the best imaginable health state
Health Status | 12 months
  Euro Qual (EQ)-Visual Analog Scale, Participants rate their perceived health status on a scale of 0-100 with 0 indicating the worst imaginable health state and 100 indicating the best imaginable health state
Health Status | 18 months
  Euro Qual (EQ)-Visual Analog Scale, Participants rate their perceived health status on a scale of 0-100 with 0 indicating the worst imaginable health state and 100 indicating the best imaginable health state
C-reactive protein (CRP) | Baseline
  CRP will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 1.33 Max 49,600
C-reactive protein | 12 months
  CRP will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 1.33 Max 49,600
Interleukin 1-Beta (IL1-beta) | Baseline
  IL1-beta will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.05 Max 375
Interleukin 1-Beta | 12 months
  IL1-beta will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.05 Max 375
Interleukin 1-Alpha (IL1-alpha) | Baseline
  IL1-alpha will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.09 Max 278
Interleukin 1-Alpha | 12 months
  IL1-alpha will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.09 Max 278
Tumor Necrosis Factor-alpha (TNF-alpha) | Baseline
  TNF-alpha will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.04 Max 248
Tumor Necrosis Factor-alpha | 12 months
  TNF-alpha will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.04 Max 248
Tumor Necrosis Factor-beta | Baseline
  TNF-beta will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.08 Max 458
Tumor Necrosis Factor-beta | 12 months
  TNF-beta will be measured from human plasma using the Mesoscale Discovery Human Biomarker Panel Unit pg/mL Min 0.08 Max 458

OTHER OUTCOMES:
Self-Efficacy | Baseline
  Barriers Self-Efficacy Scale, assessing self-efficacy or confidence in exercising behavior. 13 items rated on a 100-point scale (each statement is scored on a 100-point percentage scale with 10-point increments.) Higher score values indicated greater perceived self-efficacy.
Self-Efficacy | 6 months
  Barriers Self-Efficacy Scale, assessing self-efficacy or confidence in exercising behavior. 13 items rated on a 100-point scale (each statement is scored on a 100-point percentage scale with 10-point increments.) Higher score values indicated greater perceived self-efficacy.
Self-Efficacy | 12 months
  Barriers Self-Efficacy Scale, assessing self-efficacy or confidence in exercising behavior. 13 items rated on a 100-point scale (each statement is scored on a 100-point percentage scale with 10-point increments.) Higher score values indicated greater perceived self-efficacy.
Self-Efficacy | 18 months
  Barriers Self-Efficacy Scale, assessing self-efficacy or confidence in exercising behavior. 13 items rated on a 100-point scale (each statement is scored on a 100-point percentage scale with 10-point increments.) Higher score values indicated greater perceived self-efficacy.
Outcome Expectations | Baseline
  Multi-Dimensional Outcome Expectation for Exercise, 15-items assessed on a 5-point Likert scale from 1 (strongly disagree to 5 (strongly agree), measuring 3 domains of outcome expectations for exercise. High scores indicate a higher level of outcome expectations for exercise.
Outcome Expectations | 6 months
  Multi-Dimensional Outcome Expectation for Exercise, 15-items assessed on a 5-point Likert scale from 1 (strongly disagree to 5 (strongly agree), measuring 3 domains of outcome expectations for exercise. High scores indicate a higher level of outcome expectations for exercise.
Outcome Expectations | 12 months
  Multi-Dimensional Outcome Expectation for Exercise, 15-items assessed on a 5-point Likert scale from 1 (strongly disagree to 5 (strongly agree), measuring 3 domains of outcome expectations for exercise. High scores indicate a higher level of outcome expectations for exercise.
Outcome Expectations | 18 months
  Multi-Dimensional Outcome Expectation for Exercise, 15-items assessed on a 5-point Likert scale from 1 (strongly disagree to 5 (strongly agree), measuring 3 domains of outcome expectations for exercise. High scores indicate a higher level of outcome expectations for exercise.
Attitudes toward exercise | Baseline
  Attitudes Toward Physical Activity/Exercise Scale, 14 items assessed on a 5-point Likert scale from 1 (disagree a lot) to 5 (agree a lot), values range from 14-70 with higher scores indicating a more positive attitude.
Attitudes toward exercise | 6 months
  Attitudes Toward Physical Activity/Exercise Scale, 14 items assessed on a 5-point Likert scale from 1 (disagree a lot) to 5 (agree a lot), values range from 14-70 with higher scores indicating a more positive attitude.
Attitudes toward exercise | 12 months
  Attitudes Toward Physical Activity/Exercise Scale, 14 items assessed on a 5-point Likert scale from 1 (disagree a lot) to 5 (agree a lot), values range from 14-70 with higher scores indicating a more positive attitude.
Attitudes toward exercise | 18 months
  Attitudes Toward Physical Activity/Exercise Scale, 14 items assessed on a 5-point Likert scale from 1 (disagree a lot) to 5 (agree a lot), values range from 14-70 with higher scores indicating a more positive attitude.
Self-Regulation | Baseline
  Physical Activity Self-Regulation Scale, 12 items assessed on a 5-point Likert scale from 1 (never) to 5 (very often), scores range from 12-60, with higher scores indicating greater use of self-regulatory strategies for physical activity.
Self-Regulation | 6 months
  Physical Activity Self-Regulation Scale, 12 items assessed on a 5-point Likert scale from 1 (never) to 5 (very often), scores range from 12-60, with higher scores indicating greater use of self-regulatory strategies for physical activity.
Self-Regulation | 12 months
  Physical Activity Self-Regulation Scale, 12 items assessed on a 5-point Likert scale from 1 (never) to 5 (very often), scores range from 12-60, with higher scores indicating greater use of self-regulatory strategies for physical activity.
Self-Regulation | 18 months
  Physical Activity Self-Regulation Scale, 12 items assessed on a 5-point Likert scale from 1 (never) to 5 (very often), scores range from 12-60, with higher scores indicating greater use of self-regulatory strategies for physical activity.
Informational Support | Baseline
  PROMIS Informational Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived informational support.
Informational Support | 6 months
  PROMIS Informational Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived informational support.
Informational Support | 12 months
  PROMIS Informational Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived informational support.
Informational Support | 18 months
  PROMIS Informational Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived informational support.
Instrumental Support | Baseline
  PROMIS Instrumental Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived instrumental support.
Instrumental Support | 6 months
  PROMIS Instrumental Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived instrumental support.
Instrumental Support | 12 months
  PROMIS Instrumental Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived instrumental support.
Instrumental Support | 18 months
  PROMIS Instrumental Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating greater perceived instrumental support.
Social Isolation | Baseline
  PROMIS Social Isolation Short Form 4a, 4 items assessed on a Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating a higher perceived social isolation.
Social Isolation | 6 months
  PROMIS Social Isolation Short Form 4a, 4 items assessed on a Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating a higher perceived social isolation.
Social Isolation | 12 months
  PROMIS Social Isolation Short Form 4a, 4 items assessed on a Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating a higher perceived social isolation.
Social Isolation | 18 months
  PROMIS Social Isolation Short Form 4a, 4 items assessed on a Likert scale from 1 (never) to 5 (always) with raw scores ranging from 4-20, and higher scores indicating a higher perceived social isolation.
Emotional Support | Baseline
  PROMIS Emotional Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always), with raw scores between 4-20, and higher scores indicating greater perceived emotional support.
Emotional Support | 6 months
  PROMIS Emotional Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always), with raw scores between 4-20, and higher scores indicating greater perceived emotional support.
Emotional Support | 12 months
  PROMIS Emotional Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always), with raw scores between 4-20, and higher scores indicating greater perceived emotional support.
Emotional Support | 18 months
  PROMIS Emotional Support Short Form 4a, 4 items assessed on a 5-point Likert scale from 1 (never) to 5 (always), with raw scores between 4-20, and higher scores indicating greater perceived emotional support.
Types of Physical Activity | Baseline
  International Physical Activity Questionnaire, 4-item questionnaire, 3 of the items have 1 possible subsequent item. Answers are related to days per week and hours/minutes per day respondents perform an activity.
Types of Physical Activity | 6 months
  International Physical Activity Questionnaire, 4-item questionnaire, 3 of the items have 1 possible subsequent item. Answers are related to days per week and hours/minutes per day respondents perform an activity.
Types of Physical Activity | 12 months
  International Physical Activity Questionnaire, 4-item questionnaire, 3 of the items have 1 possible subsequent item. Answers are related to days per week and hours/minutes per day respondents perform an activity.
Types of Physical Activity | 18 months
  International Physical Activity Questionnaire, 4-item questionnaire, 3 of the items have 1 possible subsequent item. Answers are related to days per week and hours/minutes per day respondents perform an activity.
Fatigue | Baseline
  Multidimensional Fatigue Symptom Inventory - Short Form, 30 items assess on a 5-point Likert scale from 0 (not at all) to 4 (extremely), possible values range from -24-96 with higher scores indicating a higher level of fatigue.
Fatigue | 6 months
  Multidimensional Fatigue Symptom Inventory - Short Form, 30 items assess on a 5-point Likert scale from 0 (not at all) to 4 (extremely), possible values range from -24-96 with higher scores indicating a higher level of fatigue.
Fatigue | 12 months
  Multidimensional Fatigue Symptom Inventory - Short Form, 30 items assess on a 5-point Likert scale from 0 (not at all) to 4 (extremely), possible values range from -24-96 with higher scores indicating a higher level of fatigue.
Fatigue | 18 months
  Multidimensional Fatigue Symptom Inventory - Short Form, 30 items assess on a 5-point Likert scale from 0 (not at all) to 4 (extremely), possible values range from -24-96 with higher scores indicating a higher level of fatigue.
Cognitive Assessment | Baseline
  Montreal Cognitive Assessment, 12 items measuring 7 cognitive domains, scores range from 0-30, with higher scores indicating better cognitive function.
Cognitive Assessment | 6 months
  Montreal Cognitive Assessment, 12 items measuring 7 cognitive domains, scores range from 0-30, with higher scores indicating better cognitive function.
Cognitive Assessment | 12 months
  Montreal Cognitive Assessment, 12 items measuring 7 cognitive domains, scores range from 0-30, with higher scores indicating better cognitive function.
Cognitive Assessment | 18 months
  Montreal Cognitive Assessment, 12 items measuring 7 cognitive domains, scores range from 0-30, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Windy W Alonso, PhD, Principal Investigator — University of Virginia; Bunny Pozehl, PhD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in the NHLBI Data Repository under the standard procedures utilized by NHLBI to allow others access to the data. All data from baseline, months 6, 12 and 18 will be provided. Procedural-based data such as the cardiopulmonary exercise test results and the heart rate monitor data will also be provided.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available beginning 9 months after the publication of primary outcome results.
Access Criteria: Researchers that desire access to data from this study will be required to provide a methodologically sound proposal and comply with the standards outlined in the NHLBI data repository.

REFERENCES:
- [Background] Shah SJ, Borlaug BA, Kitzman DW, McCulloch AD, Blaxall BC, Agarwal R, Chirinos JA, Collins S, Deo RC, Gladwin MT, Granzier H, Hummel SL, Kass DA, Redfield MM, Sam F, Wang TJ, Desvigne-Nickens P, Adhikari BB. Research Priorities for Heart Failure With Preserved Ejection Fraction: National Heart, Lung, and Blood Institute Working Group Summary. Circulation. 2020 Mar 24;141(12):1001-1026. doi: 10.1161/CIRCULATIONAHA.119.041886. Epub 2020 Mar 23. PMID 32202936
- [Background] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Fleg JL, Cooper LS, Borlaug BA, Haykowsky MJ, Kraus WE, Levine BD, Pfeffer MA, Pina IL, Poole DC, Reeves GR, Whellan DJ, Kitzman DW; National Heart, Lung, and Blood Institute Working Group. Exercise training as therapy for heart failure: current status and future directions. Circ Heart Fail. 2015 Jan;8(1):209-20. doi: 10.1161/CIRCHEARTFAILURE.113.001420. No abstract available. PMID 25605639
- [Background] Pandey A, Parashar A, Kumbhani D, Agarwal S, Garg J, Kitzman D, Levine B, Drazner M, Berry J. Exercise training in patients with heart failure and preserved ejection fraction: meta-analysis of randomized control trials. Circ Heart Fail. 2015 Jan;8(1):33-40. doi: 10.1161/CIRCHEARTFAILURE.114.001615. Epub 2014 Nov 16. PMID 25399909
- [Background] Pozehl BJ, Duncan K, Hertzog M, McGuire R, Norman JF, Artinian NT, Keteyian SJ. Study of adherence to exercise in heart failure: the HEART camp trial protocol. BMC Cardiovasc Disord. 2014 Nov 29;14:172. doi: 10.1186/1471-2261-14-172. PMID 25433674
- [Background] Pozehl BJ, McGuire R, Duncan K, Kupzyk K, Norman J, Artinian NT, Deka P, Krueger SK, Saval MA, Keteyian SJ. Effects of the HEART Camp Trial on Adherence to Exercise in Patients With Heart Failure. J Card Fail. 2018 Oct;24(10):654-660. doi: 10.1016/j.cardfail.2018.06.007. Epub 2018 Aug 16. PMID 30010027
- [Background] Warehime S, Dinkel D, Alonso W, Pozehl B. Long-term exercise adherence in patients with heart failure: A qualitative study. Heart Lung. 2020 Nov-Dec;49(6):696-701. doi: 10.1016/j.hrtlng.2020.08.016. Epub 2020 Aug 27. PMID 32861888
- [Background] Alonso WW, Kupzyk K, Norman J, Bills SE, Bosak K, Dunn SL, Deka P, Pozehl B. Negative Attitudes, Self-efficacy, and Relapse Management Mediate Long-Term Adherence to Exercise in Patients With Heart Failure. Ann Behav Med. 2021 Oct 4;55(10):1031-1041. doi: 10.1093/abm/kaab002. PMID 33580663
- [Background] Norman JF, Kupzyk KA, Artinian NT, Keteyian SJ, Alonso WS, Bills SE, Pozehl BJ. The influence of the HEART Camp intervention on physical function, health-related quality of life, depression, anxiety and fatigue in patients with heart failure. Eur J Cardiovasc Nurs. 2020 Jan;19(1):64-73. doi: 10.1177/1474515119867444. Epub 2019 Aug 2. PMID 31373222
- [Background] Keteyian SJ. Exercise training in congestive heart failure: risks and benefits. Prog Cardiovasc Dis. 2011 May-Jun;53(6):419-28. doi: 10.1016/j.pcad.2011.02.005. PMID 21545928
- [Background] Pozehl BJ, Mcguire R, Duncan K, Hertzog M, Deka P, Norman J, Artinian NT, Saval MA, Keteyian SJ. Accelerometer-Measured Daily Activity Levels and Related Factors in Patients With Heart Failure. J Cardiovasc Nurs. 2018 Jul/Aug;33(4):329-335. doi: 10.1097/JCN.0000000000000464. PMID 29538050